CLINICAL TRIAL: NCT02184117
Title: CONTRAST (Can cONTrast Injection Better Approximate FFR compAred to Pure reSTing Physiology?)
Acronym: CONTRAST
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Nils Johnson, Associate Professor of Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0399
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve, Myocardial; Adenosine; Contrast Media
MeSH Terms: conditions — Coronary Artery Disease | interventions — Adenosine; Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Entire cohort undergoes paired testing
  Interventions: Drug: Adenosine; Drug: Contrast Media; Drug: Resting conditions

INTERVENTIONS:
Drug: Adenosine — Intracoronary or intravenous adenosine to induce hyperemia for reference FFR
Drug: Contrast Media — Intracoronary injection of contrast medium to induce hyperemia for "contrast FFR"
Drug: Resting conditions — Baseline measurement of aortic and coronary pressures

SUMMARY:
The purpose of this study is to determine the diagnostic performances of iodine contrast medium and resting conditions to predict fractional flow reserve (FFR). Reference FFR will be measured using standard adenosine. We hypothesize that contrast FFR will offer superior diagnostic agreement compared to resting conditions.

DETAILED DESCRIPTION:
We are conducting a diagnostic accuracy study. The reference standard is adenosine-derived FFR. The diagnostic tests undergoing evaluation are resting conditions and hyperemia induced by intracoronary injection of contrast medium. While all these tests give a continuous result, we will apply binary cutoffs for comparison to FFR≤0.8 as the reference standard. Subjects will be selected prospectively from consecutive patients undergoing FFR assessment for standard clinical indications. The paired comparative design means that each patient will undergo resting (baseline), post-contrast, and adenosine-derived measurements. To enhance test integrity, all pressure recordings will be analyzed in a central physiology core laboratory blinded to clinical data and recruiting site.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Undergoing FFR assessment for standard clinical indications.
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Prior coronary artery bypass grafting (CABG).
* Extremely tortuous or calcified coronary arteries precluding intracoronary physiologic measurements. Operators may exclude subtotal or similar high-grade lesions, which in their judgment may be threatened by pressure wire placement.
* Known severe left ventricular hypertrophy (septal wall thickness at echocardiography of >13 mm).
* Inability to receive adenosine (for example, severe reactive airway disease, marked hypotension, or advanced atrioventricular block without pacemaker).
* Recent (within 3 weeks prior to cardiac catheterization) ST-segment elevation myocardial infarction (STEMI) in any arterial distribution (not specifically target lesion).
* Culprit lesions (based on clinical judgment of the operator) for either STEMI or non-STEMI cannot be included.
* Severe cardiomyopathy (ejection fraction <30%).
* Renal insufficiency such that an additional 12 to 20 mL of contrast would, in the opinion of the operator, pose unwarranted risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing FFR assessment for standard clinical indications
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Agreement with binary FFR≤0.80 | Baseline
  To quantify any improvement in binary agreement from resting conditions to contrast medium injection, using adenosine-derived FFR≤0.8 as the reference standard.

SECONDARY OUTCOMES:
Binary diagnostic performance | Baseline
  To describe the diagnostic performance of resting conditions and contrast medium injection using sensitivity and specificity, positive and negative predictive value, and area under the receiver operating characteristic (ROC) curve, compared to adenosine-derived FFR≤0.8 as the reference standard.
Continuous relationship with FFR | Baseline
  To determine the relationship between adenosine-derived FFR and either resting conditions or contrast medium injection using scatter plots (correlation coefficient) and Bland-Altman analysis (bias and limits of agreement).

CONTACTS AND LOCATIONS:
Overall Officials: Nils P Johnson, MD, MS, Principal Investigator — University of Texas Medical School at Houston; William F Fearon, MD, Study Director — Stanford University
Locations (11):
- United States (2):
  - Stanford University, Palo Alto VA, Palo Alto, California
  - Integris Health, Oklahoma City, Oklahoma
- Cardiovascular Center (OLV-Ziekenhuis), Aalst, Belgium
- Hôpital Louis Pradel, Lyon, France
- University of Naples Federico II, Naples, Italy
- Catharina Hospital, Eindhoven, North Brabant, Netherlands
- Hospital Fernando Fonseca, Lisbon, Portugal
- South Korea (2):
  - Seoul National University College of Medicine, Seoul
  - Asan Medical Center, Seoul
- Södersjukhuset, Stockholm, Sweden
- Golden Jubilee National Hospital, Clydebank, United Kingdom

REFERENCES:
- [Background] De Bruyne B, Pijls NH, Barbato E, Bartunek J, Bech JW, Wijns W, Heyndrickx GR. Intracoronary and intravenous adenosine 5'-triphosphate, adenosine, papaverine, and contrast medium to assess fractional flow reserve in humans. Circulation. 2003 Apr 15;107(14):1877-83. doi: 10.1161/01.CIR.0000061950.24940.88. Epub 2003 Mar 31. PMID 12668522
- [Result] Johnson NP, Jeremias A, Zimmermann FM, Adjedj J, Witt N, Hennigan B, Koo BK, Maehara A, Matsumura M, Barbato E, Esposito G, Trimarco B, Rioufol G, Park SJ, Yang HM, Baptista SB, Chrysant GS, Leone AM, Berry C, De Bruyne B, Gould KL, Kirkeeide RL, Oldroyd KG, Pijls NHJ, Fearon WF. Continuum of Vasodilator Stress From Rest to Contrast Medium to Adenosine Hyperemia for Fractional Flow Reserve Assessment. JACC Cardiovasc Interv. 2016 Apr 25;9(8):757-767. doi: 10.1016/j.jcin.2015.12.273. PMID 27101902
- [Derived] Achim A, Johnson NP, Liblik K, Burckhardt A, Krivoshei L, Leibundgut G. Coronary steal: how many thieves are out there? Eur Heart J. 2023 Aug 7;44(30):2805-2814. doi: 10.1093/eurheartj/ehad327. PMID 37264699
- [Derived] Johnson NP, Matsuo H, Nakayama M, Eftekhari A, Kakuta T, Tanaka N, Christiansen EH, Kirkeeide RL, Gould KL. Combined Pressure and Flow Measurements to Guide Treatment of Coronary Stenoses. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1904-1913. doi: 10.1016/j.jcin.2021.07.041. PMID 34503741
- [Derived] Johnson NP, Collet C. Can FFR After Stenting Help Reduce Target Vessel Failure? JACC Cardiovasc Interv. 2021 Sep 13;14(17):1901-1903. doi: 10.1016/j.jcin.2021.08.001. No abstract available. PMID 34503740
- [Derived] Gould KL, Johnson NP, Roby AE, Nguyen T, Kirkeeide R, Haynie M, Lai D, Zhu H, Patel MB, Smalling R, Arain S, Balan P, Nguyen T, Estrera A, Sdringola S, Madjid M, Nascimbene A, Loyalka P, Kar B, Gregoric I, Safi H, McPherson D. Regional, Artery-Specific Thresholds of Quantitative Myocardial Perfusion by PET Associated with Reduced Myocardial Infarction and Death After Revascularization in Stable Coronary Artery Disease. J Nucl Med. 2019 Mar;60(3):410-417. doi: 10.2967/jnumed.118.211953. Epub 2018 Aug 16. PMID 30115688
- [Derived] Johnson NP, Kirkeeide RL, Gould KL. Same Lesion, Different Artery, Different FFR!? JACC Cardiovasc Imaging. 2019 Apr;12(4):718-721. doi: 10.1016/j.jcmg.2017.11.029. Epub 2018 Jan 17. No abstract available. PMID 29361484
- [Derived] Kobayashi Y, Johnson NP, Zimmermann FM, Witt N, Berry C, Jeremias A, Koo BK, Esposito G, Rioufol G, Park SJ, Nishi T, Choi DH, Oldroyd KG, Barbato E, Pijls NHJ, De Bruyne B, Fearon WF; CONTRAST Study Investigators. Agreement of the Resting Distal to Aortic Coronary Pressure With the Instantaneous Wave-Free Ratio. J Am Coll Cardiol. 2017 Oct 24;70(17):2105-2113. doi: 10.1016/j.jacc.2017.08.049. PMID 29050557
- [Derived] Nishi T, Johnson NP, De Bruyne B, Berry C, Gould KL, Jeremias A, Oldroyd KG, Kobayashi Y, Choi DH, Pijls NHJ, Fearon WF; CONTRAST Study Investigators. Influence of Contrast Media Dose and Osmolality on the Diagnostic Performance of Contrast Fractional Flow Reserve. Circ Cardiovasc Interv. 2017 Oct;10(10):e004985. doi: 10.1161/CIRCINTERVENTIONS.117.004985. PMID 29042397
- [Derived] Matsumura M, Johnson NP, Fearon WF, Mintz GS, Stone GW, Oldroyd KG, De Bruyne B, Pijls NHJ, Maehara A, Jeremias A. Accuracy of Fractional Flow Reserve Measurements in Clinical Practice: Observations From a Core Laboratory Analysis. JACC Cardiovasc Interv. 2017 Jul 24;10(14):1392-1401. doi: 10.1016/j.jcin.2017.03.031. PMID 28728652
- [Derived] Gargiulo G, Stabile E, Ferrone M, Barbato E, Zimmermann FM, Adjedj J, Hennigan B, Matsumura M, Johnson NP, Fearon WF, Jeremias A, Trimarco B, Esposito G; CONTRST Study Investigators. Diabetes does not impact the diagnostic performance of contrast-based fractional flow reserve: insights from the CONTRAST study. Cardiovasc Diabetol. 2017 Jan 13;16(1):7. doi: 10.1186/s12933-016-0494-2. PMID 28086778
- [Derived] Johnson NP, Gould KL, Di Carli MF, Taqueti VR. Invasive FFR and Noninvasive CFR in the Evaluation of Ischemia: What Is the Future? J Am Coll Cardiol. 2016 Jun 14;67(23):2772-2788. doi: 10.1016/j.jacc.2016.03.584. PMID 27282899
- [Derived] Gould KL, Johnson NP. Coronary Blood Flow After Acute MI: Alternative Truths. JACC Cardiovasc Interv. 2016 Mar 28;9(6):614-7. doi: 10.1016/j.jcin.2016.02.009. No abstract available. PMID 27013162
- [Derived] Gould KL, Johnson NP. Myocardial Bridges: Lessons in Clinical Coronary Pathophysiology. JACC Cardiovasc Imaging. 2015 Jun;8(6):705-9. doi: 10.1016/j.jcmg.2015.02.013. No abstract available. PMID 26068287
- [Derived] Gould KL, Johnson NP, Kaul S, Kirkeeide RL, Mintz GS, Rentrop KP, Sdringola S, Virmani R, Narula J. Patient selection for elective revascularization to reduce myocardial infarction and mortality: new lessons from randomized trials, coronary physiology, and statistics. Circ Cardiovasc Imaging. 2015 May;8(5):e003099. doi: 10.1161/CIRCIMAGING.114.003099. No abstract available. PMID 25977304